CLINICAL TRIAL: NCT05168670
Title: Safety of Tinted Soft Scleral Eye Shields When IPL is Applied Directly on Eyelids of Subjects With Dry Eye Disease Due to Meibomian Gland Dysfunction
Brief Title: Safety of Tinted Soft Scleral Eye Shields When IPL is Applied on Eyelids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lumenis Be Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUM-VBU-OPT-21-02
Record Dates: First submitted 2021-11-25; First posted 2021-12-23 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2021-11

CONDITIONS: Dry Eye Disease; Meibomian Gland Dysfunction
MeSH Terms: conditions — Dry Eye Syndromes; Meibomian Gland Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study arm (Experimental): Protection of eyes with tinted soft scleral eye shields followed by IPL administration directly on eyelids
  Interventions: Combination Product: Protection of eyes with tinted soft scleral eye shields

INTERVENTIONS:
Combination Product: Protection of eyes with tinted soft scleral eye shields — In subjects with dry eye disease due to meibomian gland dysfunction, protection of eyes with tinted soft scleral eye shields followed by IPL administration on eyelids
  Other Names: IPL adminstration on eyelids

SUMMARY:
The purpose of this study is to verify the safety of tinted soft scleral eye shields when IPL is applied directly on eyelids.

DETAILED DESCRIPTION:
Patients with dry eye disease due to meibomian gland dysfunction will be treated with one session of IPL applied directly on upper and lower eyelids, when eyes are protected with tinted soft scleral eye shields which prevent IPL from penetrating into ocular structures. Ocular structures will be examined with various tests (including: biomicroscopy, OCT and specular microscopy) at baseline and at 10 minutes after IPL, 24 hours after IPL, and 7 days after IPL. In addition, visual acuity will be measured at each of these times, and the patient will report of any visual symptoms at each of these times. The primary objective is to verify that no morphological or functional changes occur between the baseline and the 7 days follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to read, understand and sign an IC form
* 22 or older
* Self-assessed symptoms are consistent with dry eye (SPEED score ≥ 10)
* Signs of MGD, as detected in biomicroscopy
* Fitzpatrick skin type I-V
* Subject is willing to comply with all study procedures, including return to the clinic 1 day and 1 week after the first and only treatment within the scope of the study

Exclusion Criteria:

* • Fitzpatrick skin type VI

  * Ocular surgery or eyelid surgery, within 3 months prior to screening
  * Recent ocular trauma, within 3 months prior to screening
  * Pre-cancerous lesions, skin cancer or pigmented lesions in the planned treatment area
  * Severe active allergies, or other severe uncontrolled eye disorders affecting the ocular surface
  * Uncontrolled infections or uncontrolled immunosuppressive diseases
  * Subjects with ocular infections requiring the use of antibiotic treatment, within 3 months prior to screening
  * Legally blind in either eye
  * Ocular surface abnormality that may compromise corneal integrity in either eye (e.g., keratoconus, recurrent corneal erosion, corneal epithelial defect, Grade 3 corneal fluorescein staining, map dot fingerprint dystrophy, prior chemical burn)
  * Eyelid abnormalities that affect lid function in either eye, including: entropion, ectropion, tumor, blepharospasm, lagophthalmos, severe trichiasis, and severe ptosis
  * Prior history of cold sores or rashes in the perioral area or in the planned treatment area that could be stimulated by light at a wavelength of 560 nm to 1200 nm, including: Herpes simplex 1 & 2, Systemic Lupus erythematosus, and porphyria
  * Within 3 months prior to screening, use of photosensitive medication and/or herbs that may cause sensitivity to 560-1200 nm light exposure, including: Isotretinoin, Tetracycline, Doxycycline, and St. John's Wort
  * Over exposure to sun, within 4 weeks prior to screening
  * Moderate to severely compromised corneal health as assessed by corneal fluorescein staining
  * Trans-illumination defects
  * Anisocoria or pupil deformation
  * Anterior chamber inflammation
  * Media opacities (cataract, posterior capsule opacification, corneal edema, etc.) that preclude clear visualization of the anterior segment and retina
  * Any condition revealed whereby the investigator deems the subject inappropriate for this study

Ages: 22 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-01-25 (Actual)

PRIMARY OUTCOMES:
Ophthalmic morphological changes at 1 week after intervention | 1 week
  Opinion of the study investigator (yes/no) whether there was any change in ocular structures at 1 week after intervention (based on a series of tests including biomicroscopy, corneal fluorescein staining, anterior segment OCT, posterior segment OCT, and specular microscopy)

SECONDARY OUTCOMES:
Ophthalmic morphological changes at 10 minutes after intervention | 10 minutes
  Opinion of the study investigator (yes/no) whether there was any change in ocular structures at 10 minutes after intervention (based on a series of tests including biomicroscopy, corneal fluorescein staining, anterior segment OCT, posterior segment OCT, and specular microscopy)
Ophthalmic morphological changes at 24 hours after intervention | 24 hours
  Opinion of the study investigator (yes/no) whether there was any change in ocular structures at 24 hours after intervention (based on a series of tests including biomicroscopy, corneal fluorescein staining, anterior segment OCT, posterior segment OCT, and specular microscopy)
Objective functional change at 10 minutes after intervention | 10 minutes
  Change in best-corrected visual acuity (ETDRS chart) at 10 minutes after intervention
Objective functional change at 24 hours after intervention | 24 hours
  Change in best-corrected visual acuity (ETDRS chart) at 24 hours after intervention
Objective functional change at 1 week after intervention | 1 week
  Change in best-corrected visual acuity (ETDRS chart) at 1 week after intervention
Subjective functional change at 10 minutes after intervention | 10 minutes
  Change in perception of visual symptoms (Visual analog scale) at 10 minutes after intervention
Subjective functional change at 1 day after intervention | 1 day
  Change in perception of visual symptoms (Visual analog scale) at 1 day
  after intervention
Subjective functional change at 1 week after intervention | 1 week
  Change in perception of visual symptoms (Visual analog scale) at 1 week
  after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Rolando Toyos, MD, Principal Investigator — Toyos Clinic (Nashville, TN, USA)
Locations (1):
- Toyos Clinic, Nashville, Tennessee, United States